CLINICAL TRIAL: NCT00642018
Title: A Randomized Phase 2 Study of LY2181308 in Combination With Docetaxel Versus Docetaxel in Hormone Refractory Prostate Cancer
Brief Title: A Study of an Experimental Chemotherapy Combination to Treat Hormone Refractory Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10461; H8Z-MC-JACR (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-02-28; First posted 2008-03-24 (Estimated); Results first posted 2019-04-03 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-03

CONDITIONS: Prostate Cancer
Keywords: Hormone Refractory Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: Docetaxel (Active Comparator): Standard of care (SOC) docetaxel 75 mg/m² intravenously every 3 weeks and prednisone 5 mg orally twice daily continuously while receiving docetaxel therapy
  Interventions: Drug: docetaxel; Drug: Prednisone
- B: LY2181308 + Docetaxel (Experimental): LY2181308 administered with docetaxel 75 mg/m² intravenously every 3 weeks and prednisone 5 mg orally twice daily continuously while receiving docetaxel
  Interventions: Drug: docetaxel; Drug: LY2181308 sodium; Drug: Prednisone

INTERVENTIONS:
Drug: docetaxel — Docetaxel 75 milligrams per square meter (mg/m²) intravenously on Day 1 of a 21-day cycle. Patients may receive up to 10 cycles of study therapy or until progressive disease. Additional cycles may be approved by sponsor as long as the patient is benefitting from therapy.
Drug: LY2181308 sodium — LY2181308 sodium (referred to as LY2181308 throughout this record) administered weekly plus docetaxel 75 mg/m² intravenously administered every 21 days. Patients may receive up to 10 cycles of study therapy or until progressive disease. Additional cycles may be approved by sponsor as long as the patient is benefitting from therapy.
  Arms: B: LY2181308 + Docetaxel
Drug: Prednisone — Prednisone 5 mg given orally twice daily continuously while receiving docetaxel therapy

SUMMARY:
The primary purpose of this study is to determine whether LY2181308 in combination with docetaxel is safe and effective treatment for hormone refractory prostate cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate which is metastatic and/or unresectable
* Hormone refractory prostate cancer defined as progressive based by documented 2 increase Prostate specific antigen (PSA) values over a previous reference value.
* Eastern Cooperative Oncology Group (ECOG) status 0-2
* Adequate hematological functions, liver and renal functions

Exclusion Criteria:

* Known hypersensitivity to docetaxel or taxane therapy
* Documented central nervous system or leptomeningeal metastasis at time of study entry
* Had prior treatment with chemotherapy, bone-seeking radionuclides in past 6 weeks prior to enrollment, or radiotherapy involving more than 25% of marrow producing area.
* Evidence of painful and/or destructive bone metastases for which radiation therapy, bisphosphonates or bone-seeking radionuclides are necessary.
* Have received treatment in the last 30 day with a drug which has not received regulatory approval for any indication at the time of study entry.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2008-03; Primary Completion 2011-08 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM-5PM Eastern time (UTC/GMT-5 hours, EST), Study Director — Eli Lilly and Company
Locations (17):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee, United States
- Germany (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Augsburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanover
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heilbronn
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Homburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Muenchen-Planegg
- Poland (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kielce
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Olsztyn
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- Spain (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Benidorm
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elda
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pamplona

REFERENCES:
- [Derived] de Liano AG, Reig O, Mellado B, Martin C, Rull EU, Maroto JP. Prognostic and predictive value of plasma testosterone levels in patients receiving first-line chemotherapy for metastatic castrate-resistant prostate cancer. Br J Cancer. 2014 Apr 29;110(9):2201-8. doi: 10.1038/bjc.2014.189. Epub 2014 Apr 10. PMID 24722180
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Docetaxel: Docetaxel 75 milligrams per square meter (mg/m²) intravenously on Day 1 of a 21-day cycle. Prednisone 5 mg given orally twice daily continuously while receiving docetaxel therapy.
- LY2181308 + Docetaxel: LY2181308 loading dose of 750 mg intravenously on Days 1-3, followed by a maintenance dose of 750 mg on Days 8 and 15 during first 21-day cycle. LY2181308 750 mg intravenously on Days 1, 8 and 15 in combination with docetaxel 75 mg/m² on Day 1 of every 21-day cycle from Cycle 2 and beyond. Prednisone 5 mg given orally twice daily continuously while receiving docetaxel therapy.
Period: Overall Study
Arm/Group | Docetaxel | LY2181308 + Docetaxel
Started | 52 | 102
Received at Least One Dose of Study Drug | 51 | 98
Completed | 24 (Participants who completed 10 cycles of treatment.) | 23 (Participants who completed 10 cycles of treatment.)
Not Completed | 28 | 79
Not completed — Adverse Event | 11 | 36
Not completed — Withdrawal by Subject | 4 | 10
Not completed — Progressive Disease | 13 | 18
Not completed — Physician Decision | 0 | 10
Not completed — Protocol Violation | 0 | 1
Not completed — Death | 0 | 3
Not completed — Entry Criteria Not Met | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Docetaxel | LY2181308 + Docetaxel | Total
Number analyzed (Participants) | 51 | 98 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.09 (9.33) | 68.25 (8.70) | 68.20 (8.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 51 | 98 | 149
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 49 | 94 | 143
  African | 1 | 3 | 4
  Hispanic | 0 | 1 | 1
  East Asian | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 10 | 14
  Spain | 16 | 25 | 41
  Poland | 17 | 29 | 46
  Germany | 14 | 33 | 47
  Puerto Rico | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) in Participants With Hormone Refractory Prostate Cancer (HRPC) Administered LY2181308 Sodium Plus Docetaxel Compared to Docetaxel Alone
Description: PFS is defined as the time from date of first dose to the first observation of progression of disease (PD) or death due to any cause. PD was determined using the Response Evaluation Criteria In Solid Tumors (RECIST) criteria. PD is ≥20% increase in sum of longest diameter of target lesions and/or a new lesion. For participants who had no PD or death, PFS was censored at their last contact. Participants were still followed for PFS after they stopped receiving study drug.
Time Frame: Baseline to measured progressive disease or death due to any cause up to 44.68 months
Population: All randomized participants who received at least one dose of the study drug. The numbers of participants censored were 10 (Docetaxel group) and 22 (LY2181308 + Docetaxel group).
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Docetaxel | LY2181308 + Docetaxel
Number analyzed (Participants) | 51 | 98
months | 9.00 [7.00 to 10.09] | 8.64 [7.39 to 10.45]

2. Primary Outcome: Number of Participants With Adverse Events (Safety)
Description: Data are presented as number of participants who experienced serious adverse events or all other nonserious adverse events during the study including the 30-day follow-up period. A summary of serious adverse events and other nonserious adverse events is located in the Reported Adverse Event section. The participants received maximum 24 cycles of treatment (1cycle = 3 weeks). Safety data were collected up to 24 cycles plus 30 days of follow-up for a total up to 19 months.
Time Frame: First treatment dose up to 19 months
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel | LY2181308 + Docetaxel
Number analyzed (Participants) | 51 | 98
Participants
  Serious Adverse Events | 11 | 47
  Other Nonserious Adverse Events | 50 | 94

3. Secondary Outcome: Adverse Event Profile
Description: Data presented are the number of participants with all treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs), discontinuations due to SAEs and AEs, and deaths that occurred in this study that were assessed by investigators as possibly related to study drug. The participants received maximum 24 cycles of treatment (1cycle = 3 weeks). Safety data were collected up to 24 cycles plus 30 days of follow-up for a total up to 19 months.
Time Frame: First treatment dose up to 19 months
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel | LY2181308 + Docetaxel
Number analyzed (Participants) | 51 | 98
Participants
  TEAEs | 45 | 91
  SAEs | 5 | 27
  Discontinuations due to AEs | 6 | 22
  Discontinuations due to SAEs | 1 | 3
  Death | 0 | 0

4. Secondary Outcome: Pharmacokinetics of Docetaxel: Area Under the Concentration Time Curve From Time Zero to Infinity (AUC0-infinity)
Time Frame: Predose up to 8 hours postdose in Cycle 1
Population: All randomized participants who received at least one dose of the study drug and had pharmacokinetics data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*h/mL)
Arm/Group | Docetaxel | LY2181308 + Docetaxel
Number analyzed (Participants) | 24 | 48
nanograms*hour per milliliter (ng*h/mL) | 825 (56.6) | 799 (59.7)

5. Secondary Outcome: Prostate Specific Antigen (PSA) Kinetics: Percentage of Participants With PSA Response (Response Rate)
Description: PSA response was defined as a post-baseline PSA level decline of at least 50% relative to the baseline value. Response rate calculated as 100*n/N where n=the number of participants with responses and N=the total number of participants treated.
Time Frame: Baseline, 18 months
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Docetaxel | LY2181308 + Docetaxel
Number analyzed (Participants) | 51 | 98
percentage of participants | 56.9 | 56.1

6. Secondary Outcome: Estimate Overall Survival
Description: Overall survival is defined as the time from date of first treatment to the date of death due to any cause. For participants who were alive, overall survival was censored at their last contact. Participants were still followed for overall survival after they stopped receiving study drug.
Time Frame: First treatment to death due to any cause up to 45.54 months
Population: All randomized participants who received at least one dose of study drug. The numbers of participants censored were 25 (Docetaxel group) and 49 (LY2181308 + Docetaxel group).
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Docetaxel | LY2181308 + Docetaxel
Number analyzed (Participants) | 51 | 98
months | 29.04 [20.11 to 39.26] | 27.04 [19.94 to 33.41]

7. Secondary Outcome: Estimate Duration of Overall Response
Description: The duration of response [complete response (CR) or partial response (PR)] was defined as the time from first objective status assessment of CR or PR to the first time of progression or death as a result of any cause. CR or PR is classified by the investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST) guidelines. CR is disappearance of all target and non-target lesions; PR is ≥30% decrease in sum of longest diameter of target lesions. For participants who had no progression or death, the duration of response was censored at their last contact.
Time Frame: Time of response to time of measured progressive disease up to 41.00 months
Population: All randomized participants who received at least one dose of the study drug and had complete response (CR) or partial response (PR). The numbers of participants censored were 3 (Docetaxel group) and 1 (LY2181308 + Docetaxel group).
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Docetaxel | LY2181308 + Docetaxel
Number analyzed (Participants) | 11 | 10
months | 10.81 [7.49 to 14.29] | 9.66 [6.93 to 11.07]

8. Secondary Outcome: Percentage of Participants With Complete Response or Partial Response (Overall Response Rate)
Description: Overall response rate was defined as the percentage of participants who achieved a complete response (CR) or partial response (PR) per the Response Evaluation Criteria In Solid Tumors (RECIST) criteria. CR is disappearance of all target and non-target lesions; PR is ≥30% decrease in sum of longest diameter of target lesions. Objective response rate is calculated as a total number of participants with CR or PR divided by the total number of participants treated multiplied by 100.
Time Frame: Baseline to measured progressive disease up to 41.00 months
Population: All randomized participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Docetaxel | LY2181308 + Docetaxel
Number analyzed (Participants) | 51 | 98
percentage of participants | 21.6 [13 to 33] | 10.2 [6 to 17]

9. Secondary Outcome: Change From Baseline to Day 21 in Granulocyte Colony Stimulating Factor(G-CSF) (Assess Biomarker Responses)
Description: G-CSF [international units per milliliter (IU/mL)] was used to estimate biomarker responses and is presented as the percentage change from baseline.
Time Frame: Baseline, 21 days
Population: All randomized participants who received at least one dose of study drug and had G-CSF measurement at baseline and 21 days.
Measure: Number; unit: percentage change
Groups:
- LY2181308: LY2181308 loading dose of 750 mg intravenously on Days 1-3, followed by a maintenance dose of 750 mg on Days 8 and 15 during first cycle.
Arm/Group | Docetaxel | LY2181308
Number analyzed (Participants) | 49 | 98
percentage change | -32.5 | 233.3

10. Secondary Outcome: Functional Assessment of Cancer Therapy-Prostate Cancer (FACT-P) Total Score at 3 Months (Participant Reported Outcomes)
Description: The FACT-P is a 39-item participant-rated questionnaire which assesses physical well-being (7 items), social/family well-being (7 items), emotional well-being (6 items), functional well-being (7 items), and additional prostate cancer specific concerns (12 items). All items are scored from 0 (not at all) to 4 (very much). The total FACT-P score ranges from 0-156, with higher scores representing a better quality of life with fewer symptoms.
Time Frame: 3 months
Population: All randomized participants who received at least one dose of study drug and had FACT-P assessment at 3 months.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Docetaxel | LY2181308 + Docetaxel
Number analyzed (Participants) | 42 | 74
units on a scale | 117 [108 to 128] | 115 [93 to 129]

11. Secondary Outcome: Functional Assessment of Cancer Therapy-General (FACT-G) Total Score at 3 Months (Evaluate Clinical Symptoms)
Description: The total FACT-G is the sum of 4 subscale scores on the FACT-Prostate Cancer (FACT-P) participant-rated questionnaire representing general cancer symptoms: physical well-being (7 items), social/family well-being (7 items), emotional well-being (6 items), and functional well-being (7 items). All items are scored from 0 (not at all) to 4 (very much). The total FACT-G score ranges from 0-108, with higher scores representing a better quality of life with fewer symptoms.
Time Frame: 3 months
Population: All randomized participants who received at least one dose of study drug and had FACT-G assessment at 3 months.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Docetaxel | LY2181308 + Docetaxel
Number analyzed (Participants) | 42 | 75
units on a scale | 84 [75 to 92] | 80 [66 to 94]

12. Other Pre Specified Outcome: Number of Participants Who Died Due to Progressive Disease During the 30 Days Following Discontinuation From Study Treatment
Time Frame: Study treatment discontinuation up to 30 days post study treatment discontinuation
Population: All randomized participants who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel | LY2181308 + Docetaxel
Number analyzed (Participants) | 51 | 98
Participants | 1 | 0

ADVERSE EVENTS:
Description: Deaths due to progressive disease are not considered adverse events and are reported in the Other Pre-Specified outcome measure for those who died during the 30-day post study treatment follow-up period.
Arm/Group | Docetaxel | LY2181308 + Docetaxel
Serious Adverse Events (participants affected / at risk) | 11/51 | 47/98
Other Adverse Events (participants affected / at risk) | 50/51 | 94/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel (N=51) | LY2181308 + Docetaxel (N=98)
Anaemia (Blood and lymphatic system disorders) | 1 (3) | 4 (5)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 5 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (3)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1) — Resulted in 1 death in the LY2181308 + Docetaxel group.
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Deafness unilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 6 (7)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Asthenia (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 5 (5)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1)
Febrile infection (Infections and infestations) | 0 (0) | 2 (2)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3)
Sepsis (Infections and infestations) | 0 (0) | 3 (3) — Resulted in 1 death in the LY2181308 + Docetaxel group.
Septic shock (Infections and infestations) | 0 (0) | 3 (3) — Resulted in 1 death in the LY2181308 + Docetaxel group.
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cranial nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel (N=51) | LY2181308 + Docetaxel (N=98)
Anaemia (Blood and lymphatic system disorders) | 10 (21) | 39 (59)
Leukopenia (Blood and lymphatic system disorders) | 15 (51) | 34 (87)
Lymphopenia (Blood and lymphatic system disorders) | 3 (3) | 5 (5)
Neutropenia (Blood and lymphatic system disorders) | 30 (106) | 58 (172)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 47 (87)
Cushingoid (Endocrine disorders) | 3 (3) | 0 (0)
Lacrimation increased (Eye disorders) | 3 (3) | 3 (5)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 13 (17)
Abdominal pain upper (Gastrointestinal disorders) | 5 (8) | 6 (6)
Constipation (Gastrointestinal disorders) | 6 (9) | 23 (30)
Diarrhoea (Gastrointestinal disorders) | 20 (36) | 42 (84)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 14 (16)
Dyspepsia (Gastrointestinal disorders) | 5 (8) | 7 (7)
Nausea (Gastrointestinal disorders) | 13 (20) | 41 (87)
Stomatitis (Gastrointestinal disorders) | 4 (5) | 8 (10)
Vomiting (Gastrointestinal disorders) | 3 (4) | 24 (38)
Asthenia (General disorders) | 13 (26) | 21 (35)
Chest pain (General disorders) | 0 (0) | 5 (5)
Chills (General disorders) | 1 (1) | 12 (13)
Fatigue (General disorders) | 22 (44) | 38 (72)
Influenza like illness (General disorders) | 2 (2) | 9 (13)
Mucosal inflammation (General disorders) | 8 (10) | 9 (15)
Oedema peripheral (General disorders) | 11 (15) | 34 (41)
Pyrexia (General disorders) | 5 (5) | 35 (43)
Bronchitis (Infections and infestations) | 1 (1) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 4 (4)
Urinary tract infection (Infections and infestations) | 1 (2) | 6 (11)
Alanine aminotransferase increased (Investigations) | 0 (0) | 9 (17)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 8 (12)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 5 (6)
Weight decreased (Investigations) | 5 (5) | 15 (16)
Decreased appetite (Metabolism and nutrition disorders) | 11 (14) | 26 (31)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (13) | 11 (23)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 6 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (3) | 9 (10)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 6 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 15 (18)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 8 (12)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (7)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 8 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (6) | 10 (13)
Dizziness (Nervous system disorders) | 7 (8) | 10 (12)
Dysgeusia (Nervous system disorders) | 12 (20) | 26 (38)
Headache (Nervous system disorders) | 2 (2) | 13 (24)
Neuropathy peripheral (Nervous system disorders) | 4 (5) | 7 (10)
Paraesthesia (Nervous system disorders) | 7 (7) | 12 (15)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (8) | 6 (6)
Syncope (Nervous system disorders) | 2 (3) | 6 (6)
Insomnia (Psychiatric disorders) | 5 (5) | 4 (5)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 13 (14)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 21 (26)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 10 (15)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 12 (12)
Alopecia (Skin and subcutaneous tissue disorders) | 22 (23) | 40 (41)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 10 (10)
Nail disorder (Skin and subcutaneous tissue disorders) | 7 (7) | 14 (14)
Onycholysis (Skin and subcutaneous tissue disorders) | 3 (4) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 9 (12)
Flushing (Vascular disorders) | 6 (18) | 3 (5)
Hot flush (Vascular disorders) | 3 (3) | 3 (3)
Hypotension (Vascular disorders) | 4 (7) | 6 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days